CLINICAL TRIAL: NCT02586779
Title: Effectiveness of WhatsApp Messenger Usage and Other Technologises on Communication Between Consulting Physicians and the Emergency Department Staff: Randomised Double-blind Controlled Trial
Brief Title: Effectiveness of WhatsApp (a Messenger Program) Usage in Emergency Department (ED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Principal Investigator, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2015/04-11
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Communication
Keywords: Referral and consultation; emergency department; WhatsApp
MeSH Terms: conditions — Communication; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- whatsApp messages (Experimental): consultations in the experimental group will be generated with whatsApp. Patients' all radiographies, laboratory results, electrocardiographs, tomography images, wound images and/or extremity pictures will be sent to consultant physician via whatsApp.
  Interventions: Other: whatsApp
- control group (Other): consultations in the control group will be generated without whatsApp.
  Interventions: Other: without whatsApp

INTERVENTIONS:
Other: whatsApp — whatsApp application will be used for consultations.
  Arms: whatsApp messages
Other: without whatsApp — whatsApp application will be not used for consultations.
  Arms: control group

SUMMARY:
Effective communication between consulting physicians and the emergency physicians is critical for patients in the emergency department. The aim of this study was to determinate effectiveness of whatsApp usage for communication between physicians.

DETAILED DESCRIPTION:
Effective communication between consulting physicians and the emergency physicians is critical for patients in the emergency department. Many hospitals still use outdated pager systems as the foundation for clinical communication between physicians and other health care professionals. But, outdated pager systems contain some problems including long waiting-times for the return of a page, high costs, frequent interruptions, and the inability to identify the location or identity of the caller. This outdated communication technologies in healthcare can place patient safety at risk. Therefore they are no longer seen as an effective communication tool given the obvious advantages of Smart phones. WhatsApp Messenger, which is a messaging program for smart phones, is the most commonly used for communication in at present. As of September 2015, WhatsApp incorporated announced more than 900 million users. This is making it the most globally popular messaging application. WhatsApp Messenger have been started to be used for communication in healthcare. So, this study aims to trial the effect of whatsApp usage for communication between physicians.

Study Design and Setting: A prospective, randomized, double-blind, controlled, single-center, clinical trial was conducted in ED of a tertiary care university hospital with an annual census of approximately 200,000 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients who performed consultation in emergency department.
2. Patients who are consulted to a physician using whatsApp on a regular basis and who is chosen by an assistant blinded to the study.

Exclusion Criteria:

1. Patients below 18 years of age
2. Missing emergency service consultations
3. Patients with more than one consultation call
4. Consultations which do not determined the arrival duration to emergency service

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
arrival duration to emergency department | one month
  Examine consulting Physicians' arrival duration to emergency department will be obtained from consultation hours in whatsApp program.

SECONDARY OUTCOMES:
examine causes of consulting Physicians' arriving late to emergency department from data obtained by questioning of an assistant blinded to the study | one month

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gulacti, M.D., Principal Investigator — Adiyaman University of Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Johnston MJ, King D, Arora S, Behar N, Athanasiou T, Sevdalis N, Darzi A. Smartphones let surgeons know WhatsApp: an analysis of communication in emergency surgical teams. Am J Surg. 2015 Jan;209(1):45-51. doi: 10.1016/j.amjsurg.2014.08.030. Epub 2014 Oct 22. PMID 25454952